CLINICAL TRIAL: NCT00208065
Title: Evaluation of Histamine, CGRP and VIP as Biological Markers for Activation of Trigeminal and Parasympathetic Nerve Fibers in Response to "Sinus" Symptoms
Brief Title: Evaluation of Histamine, CGRP and VIP as Markers for Activation of Trigeminal and Parasympathetic Nerve Fibers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinvest (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Evaluation-Histamine,CGRP,VIP; CAPSS-321
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Migraine; Sinusitis
Keywords: migraine; biological markers; rhinosinusitis; CGRP; histamine; VIP
MeSH Terms: conditions — Migraine Disorders; Sinusitis; Rhinosinusitis | interventions — almotriptan; Pseudoephedrine

INTERVENTIONS:
Drug: almotriptan or pseudoephedrine

SUMMARY:
The primary objective of this study is to evaluate histamine, CGRP and VIP levels in saliva as biological markers for activation of trigeminal and parasympathetic nerve fibers in various clinical presentations of primary headaches compared to allergic rhinosinusitis and control populations.

DETAILED DESCRIPTION:
It has been suggested that many people with self-diagnosed or physician diagnosed "sinus" headache experience symptoms that fulfill diagnostic criteria for migraine or migrainous headache. The shared symptomatology does not differentiate these disorders."Sinus" symptoms as an early manifestation of migraine may be associated with elevated levels of CGRP suggesting peripheral trigeminal activation whereas "sinus" symptoms late in migraine may have associated elevations of VIP suggesting parasymptathetic activation. Subjects without autonomic or "sinus" symptoms will not have changes in salivatory histamine, CGRP or VIP and will have values similar to controls. Subjects with rhinosinusitis will have levels or patterns of salivatory histamine, CGRP and VIP unique from migraine subjects. If "sinus symptoms" are associated with parasympathetic activation, then there should be detectable increases in VIP early in the course of nasal symptom development and, conversely, if these symptoms associate with trigeminal activation, then increases in CGRP should be detected. Five groups of 10 subjects each will be recruited. Group A without migraine, with self-described "sinus" headache or symptoms of rhinosinusitis. Group B with chronic rhinosinusitis and no history of migraine or "sinus" headache. Group C with "sinus" headache with symptoms meeting IHS criteria for migraine and symptoms of rhinosinusitis preceding the onset of headache symptoms meeting migraine criteria. Group D with symptoms of rhinosinusitis that develop late in the course of migraine after criteria for IHS migraine are met. Group E with IHS migraine, without sinus symptoms associated with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Group A: no history or migraine, self-described sinus headache or symptoms of allergic rhinosinusitis

  * Group B: history of chronic recurrent rhinosinusitis without infection
  * Group C, D, and E: fulfill criteria for IHS migraine
  * Group C and D: fulfill protocol criteria for sinus symptoms associated with migraine
  * Group E: fulfill criteria for IHS migraine and no history of sinus symptoms
  * Age 18-65, male or female
  * Must be in good health
  * If female, postmenopausal at least 1 yr or hysterectomy or tubal ligation or be incapable of pregnancy or practice protocol listed method of contraception or have negative urine pregnancy test at Visit 1
  * Able to understand and communicate with study observer
  * Able to take oral medication and adhere to and perform study procedures
  * Able to read and comprehend written instructions and willing to complete all procedures
  * Willingness to participate by signing Informed Consent

Exclusion Criteria:

* More than 15 headache days per month

  * Pathology of the salivary glands such as sialadenitis
  * History of hypersensitivity to pseudoephedrin in subjects assigned to Group B or to any triptan-like medication in Group A, C, D, and E.
  * Subjects with diabetes, salivary gland tumors, liver disease, alcoholism, and/or neuropathy
  * Pregnant or nursing
  * Subjects with any condition that would alter the content of the saliva
  * Subjects with any condition that would interfere with the conduct of the study
  * Subjects who currently use medications contraindicated by use of almotriptan
  * Subjects who currently use anti-inflammatory medication
  * History of drug or alcohol abuse that would interfere with the study
  * Subjects who have received an investigational drug or used an investigational device within 30 days of enrollment or previously participated in CAPSS-321
  * Employees of the investigator, study center, or sponsor with direct involvement in the study as well as family members of the employees or the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Baseline histamine, CGRP and VIP levels in saliva of 5 groups of subjects (A-Control group, B-Rhinosinusitis, C-Migraine with early sinus symptoms, D-Migraine with late sinus symptoms, E-Migraine without sinus symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest, Inc.
Locations (1):
- Clinvest, Inc., Springfield, Missouri, United States